CLINICAL TRIAL: NCT04103450
Title: A Phase 3 Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Vibegron in Men With Overactive Bladder (OAB) Symptoms on Pharmacological Therapy for Benign Prostatic Hyperplasia (BPH)
Brief Title: Extension Study of Vibegron in Men With Overactive Bladder (OAB) Symptoms on Pharmacological Therapy for Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URO-901-3006; 2018-003136-72 (EudraCT Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-06

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Benign Prostatic Hyperplasia; Vibegron; Beta-3 adrenergic receptor (β3-AR); β3-AR agonist
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Intervention Model Description: Long-term extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vibegron (Experimental): Participants will receive 75 milligrams (mg) vibegron orally once daily (QD).
  Interventions: Drug: Vibegron

INTERVENTIONS:
Drug: Vibegron — oral administration
  Other Names: RVT-901; MK-4618; KRP-114V; URO-901

SUMMARY:
This study will assess the long-term safety of vibegron when dosed up to 52 weeks in men with overactive bladder (OAB) symptoms on pharmacological therapy for Benign Prostatic Hyperplasia (BPH) who previously completed treatment in Study URO-901-3005 (NCT03902080).

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed participation of the 24-week double-blind treatment period in Study URO-901-3005 (NCT03902080) and demonstrated compliance with the study procedures and study medication schedule in the opinion of the investigator.
* Participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Participant has the ability to continue to receive a stable dose of Benign Prostatic Hyperplasia (BPH) treatment with either a) alpha blocker monotherapy or b) alpha blocker +5-ARI.
* In the opinion of the investigator, the participant is able and willing to comply with the requirements of the protocol, including completing study questionnaires and the Bladder Diary.

Exclusion Criteria:

* Participant experienced any Serious Adverse Event in Study URO-901-3005 that was reported as "possibly or probably related" to study treatment by the investigator.
* Participant is using any prohibited medications
* Participant has uncontrolled hyperglycemia (defined as fasting blood glucose >150 milligrams per deciliter [mg/dL] or 8.33 millimoles per Liter [mmol/L] and/or non-fasting blood glucose >200 mg/dL or 11.1 mmol/L) based on most recent available lab results in Study URO-901-3005 or uncontrolled in the opinion of the investigator.
* Participant has uncontrolled hypertension (systolic blood pressure of ≥180 millimeters of mercury [mmHg] and/or diastolic blood pressure of ≥100 mmHg) or has a resting heart rate (by pulse) >100 beats per minute.
* Participant has systolic blood pressures ≥160 mmHg but <180 mmHg, unless deemed by the investigator as safe to proceed in this study and able to complete the study per protocol.
* Participant has current evidence of any clinically significant condition, therapy, lab abnormality, or other circumstances that might, in the opinion of the investigator, confound the results of the study, interfere with the participant's ability to comply with study procedures, or make participation in the study not in the participant's best interest.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Urovant Sciences
Locations (35):
- United States (31):
  - Private Practice, Huntsville, Alabama
  - Clinical Trials Research, Lincoln, California
  - American Institute of Research, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Northern California Research Corp, Sacramento, California
  - San Diego Clinical Trials, San Diego, California
  - Skyline Urology, Torrance, California
  - Imagine Research of Palm Beach County - Urology, Boynton Beach, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Quantum Clinical Trials, Miami, Florida
  - Urology Center Of Florida, Pompano Beach, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - DelRicht Research, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Boston Clinical Trials Inc - Urology, Boston, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beaumont Hospital Royal Oak - Urology Research, Royal Oak, Michigan
  - CentraCare Clinic - Adult & Pediatric Urology, Sartell, Minnesota
  - Poplar Bluff Urology, Poplar Bluff, Missouri
  - Adult & Pediatric Urology P.C. - Urology, Omaha, Nebraska
  - Excel Clinical Research - Internal Medicine, Las Vegas, Nevada
  - Private Practice, Las Vegas, Nevada
  - Premier Urology Group, LLC, Edison, New Jersey
  - New Jersey Urology NJU, Englewood, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Advances In Health, Inc., Houston, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Seattle Urology Research Center, Burien, Washington
- Poland (4):
  - Centrum Medyczne Linden, Krakow
  - Centrum Medyczne PROMED, Krakow
  - Medicome Sp. z o.o., Oświęcim
  - Nzoz Heureka, Piaseczno

IPD SHARING:
Plan to Share IPD: Yes
Urovant is committed to sharing patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Data requests will be reviewed and approved on the basis of scientific merit. All data provided will be anonymized according to applicable laws and regulations.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be made available within 24 months after study completion and will be accessible for a time frame appropriate for the approved proposal.
Access Criteria: Access to these clinical trial data can be requested by emailing medinfo@urovant.com and will be provided following Urovant review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 276 participants who completed Study URO-901-3005 (NCT03902080) were enrolled in Study URO-901-3006 (NCT04103450) and received at least 1 dose of open-label study drug (vibegron).
Groups:
- 52-Week Vibegron Group: Participants in Study URO-901-3005 who had been randomized to receive vibegron 75 mg once daily, orally will continue to receive same treatment in Study URO-901-3006, for an additional 28 weeks. Thus, participants will receive total 52 weeks of 75 mg vibegron treatment. No dosage adjustments were allowed.
- 28-Week Vibegron Group: Participants in Study URO-901-3005 who had been randomized to receive the placebo will receive study treatment of vibegron 75 mg once daily, orally for 28 weeks during the open label extension period. No dosage adjustments were allowed.
Period: Overall Study
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Started | 142 | 134
Completed | 126 | 124
Not Completed | 16 | 10
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set Extension (SAF-Ext) consists of all participants randomized in the parent study who: a. completed the 24-week treatment period in the parent study, and b. enrolled into, and received at least 1 dose of vibegron in, this extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group | Total
Number analyzed (Participants) | 142 | 134 | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (8.60) | 67.9 (8.17) | 67.6 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 142 | 134 | 276
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 18 | 31
  White | 127 | 112 | 239
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Serious Adverse Event, and Treatment Emergent Adverse Event (>5%)
Description: Adverse events were collected in participants from time each participant provided informed consent in parent study through Follow-up Visit (approximately 5 days after the last dose of study drug) in this extension study (URO-901-3006 [NCT03902080]). For the 28-Week Vibegron group, AEs recorded prior to initiation of vibegron (ie, while receiving placebo in the parent study) were reported as AEs in the parent study. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug. TEAE of >5% has been reported.
Time Frame: Up to Week 52
Population: SAF-Ext Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Participants
  Any SAE | 2 | 3
  Any non-SAE | 17 | 3

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters - Hematocrit, hemoglobin, platelet count, white blood cells (WBC [total and differential]), and red blood cells (RBC).
Time Frame: Up to Week 52
Population: SAF-Ext Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Chemistry Parameters
Description: Blood samples were collected for the analysis of chemistry parameters - Albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bicarbonate, calcium, chloride, creatininea, glucose (fasting or nonfasting), potassium, sodium, total bilirubin, direct bilirubin, blood urea nitrogen (BUN), and total cholesterol.
Time Frame: Up to Week 52
Population: SAF-Ext Population
Measure: Count of Participants; unit: Participants
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Urinary Parameters
Description: Urine samples were collected for the analysis of urinary parameters- Blood, glucose, protein, specific gravity, microscopic exam (RBCs, WBCs, epithelial cells, and bacteria), potential of hydrogen (pH) and color
Time Frame: Up to Week 52
Population: SAF Ext Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Coagulation Parameter
Description: Blood samples were collected for the analysis of coagulation parameters- international normalized ratio (INR), prothrombin time (PT) and activated partial thromboplastin time (APTT).
Time Frame: Up to Week 52
Population: SAF Ext Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Participants | 0 | 0

6. Primary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Blood pressure measurements were taken with the participant in the sitting position. Baseline is defined as the last recorded value on or prior to the date of randomization in the parent study URO-901-3005. Change from Baseline was calculated as maximum post-Baseline value minus Baseline value.
Time Frame: Baseline; Week 52
Population: SAF-Ext Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Millimeters of mercury
  SBP | -1.2 (12.50) | 0.1 (9.31)
  DBP | 0.2 (8.79) | 1.1 (6.82)

7. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart Rate was measured with the participant in the sitting position. Baseline is defined as the last recorded value on or prior to the date of randomization in the parent study URO-901-3005. CFB was calculated as maximum post-Baseline value minus Baseline value.
Time Frame: Baseline; Week 52
Population: SAF Ext Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
Number analyzed (Participants) | 142 | 134
Beats per minute | 3.3 (9.24) | -0.7 (7.98)

8. Secondary Outcome: Change From Baseline at Week 52 in the Average Number of Micturition Episodes Per Day
Description: Micturition is defined as "Urinated in Toilet" as indicated on Bladder Diary. Micturition episodes are the number of times participants voided in the toilet as indicated on the Bladder Diary, either by marking the 'urinated in toilet' question as yes or recording non-zero volume voided. Average number of micturition episodes/day was calculated using records within the diary analysis visit divided by non-missing diary days (diary days with at least one void reported). A "Diary Day" is defined as the time between when the participants gets up for the day (ie, the time the participant got up for the day yesterday to the time participant got up for the day today; approximately a 24-hour period). The last recorded value on or prior to the date of randomization in the parent study URO-901-3005 is defined as Baseline. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline; Week 52
Population: Full Analysis Set Extension (FAS-Ext) comprises of all OAB participants who took at least one dose of vibegron in the extension study and have at least one evaluable change from Baseline micturition measurement in this study. Note that the 28-week vibegron group is not included in the change from baseline at Week 52 outcome analyses because this group receieved study treatment for 28 weeks only and no data is avaliable to report at 52 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Micturition Episodes per Day
Arm/Group | 52-Week Vibegron Group
Number analyzed (Participants) | 119
Micturition Episodes per Day | -2.43 (0.299)

9. Secondary Outcome: Change From Baseline at Week 52 in the Average Number of Urgency Episodes Per Day
Description: The number of urgency episodes was defined as the number of times a participant checked that they had the need to urinate immediately as indicated on the Bladder Diary. Average number of daily urgency episodes at each study visit was calculated as the total number of urgency episodes using records within the diary analysis visit windows divided by non-missing diary days. The last recorded value on or prior to the date of randomization in the parent study URO-901-3005 is defined as Baseline. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline; Week 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Urgency Episodes per Day
Arm/Group | 52-Week Vibegron Group
Number analyzed (Participants) | 119
Urgency Episodes per Day | -2.90 (0.422)

10. Secondary Outcome: Change From Baseline at Week 52 in the Average Number of Nocturia Episodes Per Night
Description: A nocturia episode is defined as waking to pass urine during the main sleep period as indicated on the Bladder diary. Average number of nocturia episode at each study visit was calculated as the total number of nocturia episode recorded within the diary analysis visit windows divided by non-missing diary days. The last recorded value on or prior to the date of randomization in the parent study URO-901-3005 is defined as Baseline. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline; Week 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Nocturia Episodes per Night
Arm/Group | 52-Week Vibegron Group
Number analyzed (Participants) | 119
Nocturia Episodes per Night | -1.01 (0.144)

11. Secondary Outcome: Change From Baseline at Week 52 in the Average Number of Urge Urinary Incontinence (UUI) Episodes Per Day in Participants With Incontinence
Description: The number of UUI episodes was defined as the number of times a participant checked that they had "urge" as the main reason for leakage. Average UUI episodes per day at each study visit was calculated as total number of UUI episodes within the diary analysis visit windows divided by non-missing diary days. The UUI was analyzed for participants with UI at Baseline. The last recorded value on or prior to the date of randomization in the parent study URO-901-3005 is defined as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: UUI Episodes per day
Arm/Group | 52-Week Vibegron Group
Number analyzed (Participants) | 31
UUI Episodes per day | -0.75 (0.773)

12. Secondary Outcome: Change From Baseline at Week 52 in the Average of the International Prostate Symptom Score (IPSS) Storage Score (1-week Recall)
Description: The International Prostate Symptom Score (IPSS) is a rating scale for severity of lower urinary tract symptoms (LUTS). The IPSS is based on 7 questions concerning urinary symptoms and 1 question concerning quality of life. Each question concerning urinary symptoms allows the participant to choose 1 out of 6 answers indicating increasing severity of the symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Higher scores represent greater severity of symptoms. The last recorded value on or prior to the date of randomization in the parent study URO-901-3005 is defined as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 52-Week Vibegron Group
Number analyzed (Participants) | 127
Scores on a scale | -3.5 (0.31)

13. Secondary Outcome: Change From Baseline at Week 52 in the Average Volume Voided Per Micturition
Description: Total volume voided was calculated using all urinary volumes collected regardless of whether participant checked "Urinated in Toilet" or not. Average volume voided per micturition at each study visit was calculated as the total volume voided recorded divided by the number of micturitions with volume recorded. The last recorded value on or prior to the date of randomization in the parent study URO-901-3005 is defined as Baseline. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Milliliters
Arm/Group | 52-Week Vibegron Group
Number analyzed (Participants) | 118
Milliliters | 20.56 (6.750)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: SAEs and TEAEs were collected in Safety analysis set.
Arm/Group | 52-Week Vibegron Group | 28-Week Vibegron Group
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/134
Serious Adverse Events (participants affected / at risk) | 2/142 | 3/134
Other Adverse Events (participants affected / at risk) | 17/142 | 3/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 52-Week Vibegron Group (N=142) | 28-Week Vibegron Group (N=134)
Angina pectoris (Cardiac disorders) | 1 (1) | 0
Chest pain (General disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 52-Week Vibegron Group (N=142) | 28-Week Vibegron Group (N=134)
COVID-19 (Infections and infestations) | 8 (8) | 3 (3)
Hypertension (Investigations) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor does not object to publication by Institution or Principal Investigator (PI) of results of the Trial based on information collected or generated by the Institution or PI. However, the Institution and PI are required to provide the Sponsor with an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed to ensure against any inadvertent disclosure of Sponsor Confidential Information or unprotected Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04103450/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04103450/SAP_001.pdf